CLINICAL TRIAL: NCT05750004
Title: The Deviation Between the Planned and Actual Positions of Immediate Implants Placed in the Anterior Maxilla Using the Virtual Safe Angle Concept and a Novel Computer-guided Drilling Protocol. A Prospective Clinical Trial
Brief Title: Deviation Between Virtual and Actual Computer Guided Immediate Implants Using the New Safe Angle Position Concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Abo El Futtouh (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor-Investigator, Ahmed Abo El Futtouh, Clinical director of implant speciality program, Misr International University
Organization: Misr International University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSA3231001
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Immediate Implants
Keywords: Immediate implant placement; computer guided; safe angle position; Angular deviation

STUDY DESIGN:
Intervention Model Description: A prospective clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer guided immediate implant placement (Experimental): Atraumatic extraction followed by immediate implant placement using safe angle position computer guided surgical stents.
  Interventions: Procedure: computer guided immediate implant placement

INTERVENTIONS:
Procedure: computer guided immediate implant placement — Atraumatic extraction followed by immediate implant placement using safe angle position computer guided surgical stents, followed by customized healing abutments. after 3 months, Impressions for final prosthesis will be done

SUMMARY:
The goal of this case series study is to assess the degree of angular deviation between virtual and actual computer guided immediate implant placement in anterior maxilla using the new safe angle position concept and the resultant effects on soft and hard tissues. Patients with non-restorable anterior maxillary teeth will be managed with flapless computer guided immediate implant placement fabricated using safe angle concept.

DETAILED DESCRIPTION:
Various research investigated the distance deviations at the entrance and apical points of angular deviation to investigate the clinical accuracy of implant placement using these surgical procedures. Additionally, the 3D variations between the intended and postoperative implant placements are evaluated in the mesio-distal, bucco-lingual, and vertical directions. The vertical orientations are all constrained by bone volume; nevertheless, the greatest contributors to 3D deviations in implant location are bucco-lingual and mesio-distal deviations. Few research have been done to examine the variables affecting implant placement accuracy using free-hand surgical procedures. Due to drilling errors caused by drills travelling along the paths of least resistance during IIP and socket morphology, implants frequently end up in the facial region even when surgical guidelines are present. This is more typical for anterior maxilla implants. The incisal long axis, which is perpendicular to the palate or the occlusal plane, and the root's long axis connect at an angle. The incisal plane line will be at the cingulum position or slightly palatal to it when this relation is shifted more palatally, and this position is known as the safe angle position. According to the amount of palatal bone present, the occlusion with the opposing dentition, and the type of restoration, the more palatal relocation to the cingulum is carried out. Immediate implants in the safe angle position are more likely to predictably achieve good implant location (less angular deviation), improved aesthetics and emergence profile, and less stresses on the implant.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 20 years to 50 years of both genders and in good general health.
2. Maxillary anterior tooth that cannot be retained due to non-periodontitis, including fracture, endodontic failure, and root resorption, bounded by natural teeth.
3. Intact buccal bone plate (via CBCT).
4. The extraction socket has at least 3-5 mm apical bone.

Exclusion Criteria:

* 1. Smokers 2. Pregnant and lactating females: Pregnancy as this will limit recording the outcome data eg: CBCT.

  3. Medically compromised patients, as uncontrolled diabetic patients, patients taking bisphosphonates injection for treatment of osteoporosis, patients with active cardiac diseases, patients undergoing radiotherapy or chemotherapy, or any other medical and general contraindications for the surgical procedure (i.e. ASA score ≥III) (31) 4. Patients with active infection related at the site of implant/bone graft placement.

  5. Patients with untreated active periodontal diseases. 6. Patients with parafunctional habits. 7. Refuse to participate in this study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Angular deviations | 9 months
  Angular discrepancy (measured in degrees) be-tween the planned and actual implant position respective to the center of the implant body. It is primarily ascribed to a variation in point of implant entry

CONTACTS AND LOCATIONS:
Locations (1):
- International Dental Contining Education Centre (IDCE), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No